CLINICAL TRIAL: NCT02740023
Title: Quality Control of CE-Certified Phonak Hearing Aids
Brief Title: Quality Control of CE-Certified Phonak Hearing Aids - 2015_03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Sonova2015_03
Record Dates: First submitted 2016-03-31; First posted 2016-04-15 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phonak Audéo V90-13 (Active Comparator): The Phonak Audéo V90-13 will be fitted to the participants individual hearing loss.
  Interventions: Device: Hearing Aid (Phonak Audéo V90-13)
- Successor of Phonak Audéo V90-13 (Experimental): The successor of Phonak Audéo V90-13 will be fitted to the participants individual hearing loss.
  Interventions: Device: Hearing Aid (Successor of Phonak Audéo V90-13)

INTERVENTIONS:
Device: Hearing Aid (Phonak Audéo V90-13) — Phonak's Receiver-In-the-Canal (RIC) hearing aid Audéo V90-13 will be fitted to the participants individual Hearing loss.
  Arms: Phonak Audéo V90-13
Device: Hearing Aid (Successor of Phonak Audéo V90-13) — The successor of Phonak's Receiver-In-the-Canal (RIC) hearing aid Audéo V90-13 will be fitted to the participants individual Hearing loss.
  Arms: Successor of Phonak Audéo V90-13

SUMMARY:
Phonak Hearing Systems pass through different development and study stages. At an early stage, feasibility studies are conducted to investigate new algorithms, features and functions in an isolated manner.

ELIGIBILITY:
Inclusion Criteria:

* Adult hearing impaired persons (minimum age: 18 years) with and without (experience with) hearing aids
* Good written and spoken (Swiss) German language skills
* Healthy outer ear
* Ability to fill in a questionnaire (p/eCRF) conscientiously
* Informed Consent as documented by signature

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* Inability to produce a reliable hearing test result
* Massively limited dexterity
* Known psychological problems
* Central hearing disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Speech intelligibility in percent in a quiet listening situation | One week
  The data, serving as primary outcomes are collected in a series of lab appointments. The speech intelligibility in quiet will be assessed with the aid of the german rhyme test "Einsilber-Reimtest nach von Wallenberg und Kollmeier" (WaKo). The result is the speech intelligibility in percent. Descriptive statistics will be executed in the form of determining the median and quartiles. Interference statistics will be executed by applying the appropriate parametric or non-parametric test, depending on the data's distribution. A significance level of 5% is pursued.

SECONDARY OUTCOMES:
Speech intelligibility in percent in a noisy listening situation | One week
  The data, serving as secondary outcomes are collected in a series of lab appointments. The speech intelligibility in noise will be assessed with the aid of the german rhyme test "Einsilber-Reimtest nach von Wallenberg und Kollmeier" (WaKo). The result is the speech intelligibility in percent. Descriptive statistics will be executed in the form of determining the median and quartiles. Interference statistics will be executed by applying the appropriate parametric or non-parametric test, depending on the data's distribution. A significance level of 5% is pursued.

OTHER OUTCOMES:
Initial first fit acceptance (pre-calulation) in lab | One week
  The data, serving other pre-specified outcomes are collected within the first lab appointment. The acceptance of the initial first fit will be assessed with the aid of quantitative questions within an interview. The results are points on a scale and open ended (e.g. Question: Please rate the sound quality; Answer scale: bad, poor, fair, good, excellent) . Descriptive statistics will be executed in the form of determining number of answers. Interference statistics will be executed by applying the appropriate parametric or non-parametric test, depending on the data's distribution. A significance level of 5% is pursued.
Sound quality and listening effort ratings in lab | Four weeks
  The data, serving other pre-specified outcomes are collected within the lab appointments. The sound quality and listening effort ratings will be assessed with the aid of the Multi-Stimulus Test with Hidden Reference and Anchor (MUSHRA). The results are quantitative sound quality and listening effort ratings. Descriptive statistics will be executed in the form of determining the median and quartiles. Interference statistics will be executed by applying the appropriate parametric or non-parametric test, depending on the data's distribution. A significance level of 5% is pursued.

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No